CLINICAL TRIAL: NCT03211468
Title: Effectiveness of an Intervention Program to Improve Body Image and Self-Esteem Among Female Adolescent Aesthetic Athletes.
Brief Title: Intervention Program to Improve Body Image and Self-Esteem Among Female Athletes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Tel Hai College
Record Dates: First submitted 2017-05-07; First posted 2017-07-07 (Actual); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Feeding and Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Program (Experimental): Clinical intervention designed to prevent eating disorders and promote healthy eating habits and body image among female adolescent athletes. The intervention program will include 10 45-min interactive sessions led by the researcher. Each session will include a brief theoretical background, experiential activities (artistic or cognitive / emotional) and group discussions.
  Interventions: Behavioral: Clinical intervention program to prevent eating disorders
- Control Group (No Intervention): No participation in intervention program.

INTERVENTIONS:
Behavioral: Clinical intervention program to prevent eating disorders — See previous
  Arms: Intervention Program

SUMMARY:
A controlled, randomized clinical intervention study which includes the development and activation of an intervention program designed to prevent eating disorders among adolescent female aesthetic athletes. Our hypothesis is that the intervention program will yield improvement in the participants' eating behaviors, drive for thinness, and body image as compared with the age matched control group. Results will be measured using the study questionnaire, to be filled out by the participants before, after, and three months after the completion of the program. The Questionnaire will include validated questionnaires with good psychometric qualities.

DETAILED DESCRIPTION:
Eating disorders can cause a decrease in athletic performance and affect the overall health of athletes. Athletes are exposed to an increased risk of developing pathological eating behaviors and dissatisfaction with their bodies. A number of studies have found higher rates of eating pathologies in aesthetic sports such as dance, ice skating, and gymnastics. Other studies have found that intervention programs designed to prevent eating disorders in athletes have yielded promising results. The current study will examine the effects of a controlled clinical intervention program designed to prevent eating disorders and improve the body image of female adolescent figure skaters and dancers. The program will consist of ten 45-minute interactive sessions led by the researcher. Each session will include a brief theoretical background, experiential activities (artistic or cognitive / emotional) and group discussions. The control group shall include age matched athletes who will not participate in the intervention program. The impact of the intervention shall be assessed with a nonrandomized, controlled experimental group design. To assess the impact and outcome of the intervention, all participants in the research and control groups will be asked to complete the study questionnaire at pre, post, and 3-month (after post) follow-up assessments. Process evaluation, which assesses program dissemination, attendance and relapse rates, as well as assessment of participants' satisfaction, will be performed at the end of the program. The study questionnaire includes: Personal and Demographic Information, EDI-2 (Eating Disorders Inventory), Body Esteem Scale-Mendelson, SATAQ-4 (Sociocultural Attitudes Towards Appearance Questionnaire-4), EDE-Q 8 (Eating Disorder Examination Questionnaire- 8), BAS (Body Appreciation Scale). All questionnaires have good psychometric properties. The study hypothesis is that the intervention program will result in improvement in the intervention group in terms of: disturbed eating behaviors, pursuit of thinness, body-dissatisfaction and external influences on body image compared with an age-matched control group that did not participate in the program.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 10-16
* Athletes in aesthetic sports: figure skaters, dancers and gymnasts.

Exclusion Criteria:

* Males
* Females under age 10 or over 16
* Athletes from non-aesthetic sports
* Non-athletes.

Ages: 10 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 95 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change in results of study questionnaire. | Each participant shall be assessed for a total duration of 6 months.
  Questionnaire shall be answered by study participants by hand or using Qualtrics online software. 3 points of assessment for each participant: baseline, post-intervention, and 3 months follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic College of Tel Hai, Kiryat Shmona, North of Israel, Israel

IPD SHARING:
Plan to Share IPD: No